CLINICAL TRIAL: NCT00005371
Title: Epidemiology of Acute Phase Protein and CHD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4262; R01HL049872 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Atherosclerosis

SUMMARY:
To use the Multiple Risk Factor Intervention Trial (MRFIT) stored serum bank to do nested case-control studies of various serum risk factors in coronary heart disease incidence and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

The use of stored serum from the MRFIT cohort contributed additional information on how various lipid fractions and other serum constituents interact to produce atherosclerotic disease. The cost of performing such studies on a new cohort would be many times greater.

DESIGN NARRATIVE:

The case-control study evaluated: 1) the relationship between acute phase reactants, albumin, alpha 1 glycoprotein c-reactive protein and sialic acid; 2) oxidized low density lipoprotein cholesterol (LDLC) measured by thiobarbituric acid reactive substances (TBARS), and risk of myocardial infarction or coronary heart disease death; 3) Lp(a); 4) antioxidized vitamin E and carotene. The study was done in one year because of the need to analyze the specimens shortly after they were thawed. The statistical analysis was done in collaboration with University of Minnesota Coordinating Center.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-04; Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Kuller — University of Pittsburgh